CLINICAL TRIAL: NCT03106350
Title: Symptoms Experienced and Quality of Life in Patients With Breast Cancer Receiving Radiotherapy Across One Year
Brief Title: Symptoms Experienced and Quality of Life in Breast Cancer Receiving Radiotherapy
Status: Completed | Type: Observational
Sponsor: Chulabhorn Cancer Center (Other)
Responsible Party: Principal Investigator, Saengrawee Thanthong, Principal Investigator, Chulabhorn Cancer Center
Other Study IDs: 13/2557
Record Dates: First submitted 2017-03-29; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Quality of Life
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- questionnaire: EORTC-QLQ-30 questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients. It is a copyrighted instrument, which has been translated and validated in over 100 languages and is used in more than 3,000 studies worldwide.
  Other Names: EORTC-QLQ-30 Questionnaire

SUMMARY:
EORTC-QLQ-30 questionnaire filled in by participants 6 times

DETAILED DESCRIPTION:
EORTC-QLQ-30 questionnaire filled in by participants 6 times

* 1st before receive radiotherapy
* 2nd after receive radiotherapy
* 3th 1 month after receive radiotherapy
* 4th 3 month after receive radiotherapy
* 5th 6 month after receive radiotherapy
* 6th 1 year after receive radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* good consciousness
* ability to understand and provide information
* no hearing impairment
* Eastern Cooperative Oncology Group performance level of 0 to 2

Exclusion Criteria:

* prior radiotherapy

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
symptoms experienced | Change from Baseline symptoms experienced at 1 month,3 month,6 month,1 year after radiotherapy
  symptoms experienced collected by EORTC-QLQ-30

SECONDARY OUTCOMES:
quality of life | Change from Baseline quality of life at 1 month,3 month,6 month,1 year after radiotherapy
  quality of life collected by EORTC-QLQ-30

CONTACTS AND LOCATIONS:
Overall Officials: Saengrawee Thanthong, M.N.S, Principal Investigator — Chulabhorn Hospital

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Jim HS, Andrykowski MA, Munster PN, Jacobsen PB. Physical symptoms/side effects during breast cancer treatment predict posttreatment distress. Ann Behav Med. 2007 Oct;34(2):200-8. doi: 10.1007/BF02872674. PMID 17927558
- [Background] Manning-Walsh J. Social support as a mediator between symptom distress and quality of life in women with breast cancer. J Obstet Gynecol Neonatal Nurs. 2005 Jul-Aug;34(4):482-93. doi: 10.1177/0884217505278310. PMID 16020416
- [Background] Williams SA, Schreier AM. The effect of education in managing side effects in women receiving chemotherapy for treatment of breast cancer. Oncol Nurs Forum. 2004 Jan-Feb;31(1):E16-23. doi: 10.1188/04.ONF.E16-E23. PMID 14722602
- [Background] Sahin ZA, Tan M. Quality of Life and Symptom Experience of Breast Cancer Patients Undergoing Chemotherapy. Holist Nurs Pract. 2016 Jul-Aug;30(4):193-200. doi: 10.1097/HNP.0000000000000157. PMID 27309408
- [Background] Deshields TL, Potter P, Olsen S, Liu J. The persistence of symptom burden: symptom experience and quality of life of cancer patients across one year. Support Care Cancer. 2014 Apr;22(4):1089-96. doi: 10.1007/s00520-013-2049-3. Epub 2013 Dec 3. PMID 24292095
- [Background] Roiland RA, Heidrich SM. Symptom clusters and quality of life in older adult breast cancer survivors. Oncol Nurs Forum. 2011 Nov;38(6):672-80. doi: 10.1188/11.ONF.672-680. PMID 22037330
- [Background] Liang SY, Chao TC, Tseng LM, Tsay SL, Lin KC, Tung HH. Symptom-Management Self-efficacy Mediates the Effects of Symptom Distress on the Quality of Life Among Taiwanese Oncology Outpatients With Breast Cancer. Cancer Nurs. 2016 Jan-Feb;39(1):67-73. doi: 10.1097/NCC.0000000000000244. PMID 25730592
- [Background] Wu HS, Harden JK. Symptom burden and quality of life in survivorship: a review of the literature. Cancer Nurs. 2015 Jan-Feb;38(1):E29-54. doi: 10.1097/NCC.0000000000000135. PMID 24831042
- [Background] Reed E, Kossler I, Hawthorn J. Quality of life assessments in advanced breast cancer: should there be more consistency? Eur J Cancer Care (Engl). 2012 Sep;21(5):565-80. doi: 10.1111/j.1365-2354.2012.01370.x. Epub 2012 Jun 4. PMID 22672416
- See also: 2.1. Globocan 2012: Estimate Cancer Incidence, Mortality and Prevalence Worldwide in 2012 — http://globocan.iarc.fr/Pages/fact_sheets_cancer.aspx